CLINICAL TRIAL: NCT04263246
Title: Does Medium-Term Supplementation With PhytoDyNAmic Affect Exercise Performance and Antioxidant Status in Healthy Men and Women: A Randomized Controlled Trial?
Brief Title: Medium-Term Supplementation With Herbal Extract for Exercise Performance and Antioxidant Status
Acronym: PhytoDyNAmic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 320-PDY/2019
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Exercise Performance
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PhytoDyNAmic (Experimental): Six capsules per day b.i.d.
  Interventions: Dietary Supplement: PhytoDyNAmic
- Inulin (Placebo Comparator): Six capsules per day b.i.d.
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: PhytoDyNAmic — PhytoDyNAmic (6 capsules per day)
  Arms: PhytoDyNAmic
Dietary Supplement: Inulin — Inulin (6 capsules per day)
  Arms: Inulin

SUMMARY:
We evaluated here the effects of 6-week intervention with herbal supplement on exercise performance outcomes and serum biomarkers of antioxidant status. In addition, we also assessed the long-term effects (6-month) of the intervention in elderly adults.

DETAILED DESCRIPTION:
Experimental protocol

* Double-blind, randomized, placebo-controlled cross-over trial
* 6-week intervention trial (with additiional follow-up arm after 6 months)
* Experimental intervention (PhytoDyNAmic) = 6 capsules per day
* Placebo (inulin) = 1 g per day b.i.d.
* Administration = 3 capsules with breakfast and 3 capsules with dinner
* Wash-out period = 2 weeks
* No changes in physical activity patterns and diet during the study

Outcomes assessed at baseline and at each follow-up:

* Exercise performance during incremental running-to-exhaustion test
* Serum biomarkers of antioxidant status
* Total antioxidant capacity (TAC)
* Superoxide dismutase (SOD)
* Telomerase activity

Early termination criteria

- Serious subjective side effects of an intervention (e.g. nausea, vomiting, bloating)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body mass index 19 - 25 kg/m2
* Free of major chronic diseases or acute disorders

Exclusion Criteria:

* Use of dietary supplements within 4 weeks before study commences
* Unwillingness to return for follow-up analysis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in time to exhaustion | Baseline vs. 6 weeks post-intervention
  Baseline vs. 6 weeks

SECONDARY OUTCOMES:
Change in serum superoxide dismutase | Baseline vs. 6 weeks post-intervention
  Baseline vs. 6 weeks
Change in serum total antioxidant capacity | Baseline vs. 6 weeks post-intervention
  Baseline vs. 6 weeks
Change in serum telomerase activity | Baseline vs. 6 weeks post-intervention
  Baseline vs. 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nebojsa Maksimovic, PhD, Study Chair — Faculty of Sport and PE
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No